CLINICAL TRIAL: NCT01070966
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of VYTORIN in Usual Practice
Brief Title: Vytorin Reexamination Study (0653A-174)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0653A-174; 2010_010
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: Atherosclerosis
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- VYTORIN® 10/10 (ezetimibe 10 mg/simvastatin 10 mg tablets): Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with VYTORIN® 10/10 (ezetimibe 10 mg/simvastatin 10 mg tablets)
- VYTORIN® 10/20 (ezetimibe 10 mg/simvastatin 20 mg tablets): Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with VYTORIN® 10/20 (ezetimibe 10 mg/simvastatin 20 mg tablets)
- VYTORIN® 10/40 (ezetimibe 10 mg/simvastatin 40 mg tablets): Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with VYTORIN® 10/40 (ezetimibe 10 mg/simvastatin 40 mg tablets)
- VYTORIN® 10/80 (ezetimibe 10 mg/simvastatin 80 mg tablets): Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with VYTORIN® 10/80 (ezetimibe 10 mg/simvastatin 80 mg tablets)

SUMMARY:
This survey is conducted for preparing application material for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of VYTORIN through collecting the safety and efficacy information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants Who Receives Vytorin In Usual Medical Practice Within Local Label For The First Time

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Primary Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with Vytorin
Sampling Method: Probability Sample
Enrollment: 2089 (Actual)
Dates: Start 2005-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- VYTORIN® 10/10 mg/Day to 10/80 mg/Day: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH)treated with VYTORIN® dosages ranging from 10/10(ezetimibe 10 mg/simvastatin 10 mg tablets)a day to 10/80(ezetimibe 10 mg/simvastatin 80 mg tablets)a day.
Period: Participants for Safety Evaluation
Arm/Group | VYTORIN® 10/10 mg/Day to 10/80 mg/Day
Started | 2089
Completed | 2011
Not Completed | 78
Not completed — Violation of inclusion criteria | 59
Not completed — Off-label use | 9
Not completed — Duplicate Participants | 4
Not completed — Violation inclusion criteria/off label | 3
Not completed — TMT given before date of contract | 3
Period: Participants for Efficacy Evaluation
Arm/Group | VYTORIN® 10/10 mg/Day to 10/80 mg/Day
Started | 2011
Completed | 1929
Not Completed | 82
Not completed — Lack of tmt period (<28 days) | 61
Not completed — No efficacy evaluation | 19
Not completed — Efficacy evaluation window violation | 2

BASELINE CHARACTERISTICS:
Groups:
- VYTORIN® 10/10 mg/Day to 10/80 mg/Day: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia (HoFH) treated with VYTORIN® ranging from 10/10 mg/day through 10/80 mg/day for Years 1 to 6.
Arm/Group | VYTORIN® 10/10 mg/Day to 10/80 mg/Day
Number analyzed (Participants) | 2011
Age, Customized [Number; unit: Participants]
  10 ≤age <20 | 5
  20 ≤age <30 | 22
  30 ≤age <40 | 111
  40 ≤age <50 | 391
  50 ≤age <60 | 598
  60 ≤age <70 | 600
  70 ≤age <80 | 256
  80 ≤age <90 | 28
Sex/Gender, Customized [Number; unit: participants]
  Male | 930
  Female | 1081

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Clinical and/or Laboratory Adverse Experiences While Taking VYTORIN® Within 14 Days After Treatment Discontinuation
Description: Participants who recieved VYTORIN and experienced any adverse event related or unrelated to VYTORIN®, within 14 days after treatment.
Time Frame: Up to 14 days after the treatment discontinuation
Measure: Number; unit: Percentage of Participants
Groups:
- Participants Treated With VYTORIN: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Years 1 to 6.
Arm/Group | Participants Treated With VYTORIN
Number analyzed (Participants) | 2011
Percentage of Participants | 5.72

2. Primary Outcome: Mean Percent Change From Baseline to Treatment in Lipid Parameters
Description: The mean percent change from baseline to treatment in lipid parameters (total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides[TG]) and overall efficacy was evaluated by the investigator to show if there was any(improved, unchanged, worsened) lipid parameters over a period of approximately 5 years.
Time Frame: Baseline and up to 5 years
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Participants Baseline Lipid Parameters: Participants baseline lipid parameters for Total Cholesterol, HDL cholesterol, LDL cholesterol and Triglyceride.
- Participants Treatment Lipid Parameters: Participants treatment lipid parameters for Total Cholesterol, HDL cholesterol, LDL cholesterol and Triglyceride.
Arm/Group | Participants Baseline Lipid Parameters | Participants Treatment Lipid Parameters | Participants Percent Change
Number analyzed (Participants) | 2011 | 2011 | 2011
percentage change
  TC (n = 1965, 1993, 1956) | 231.31 (46.33) | 173.00 (40.78) | -23.90 (17.45)
  HDL (n = 1805, 1782, 1705) | 49.64 (13.42) | 49.85 (13.17) | 2.06 (15.27)
  LDL (n = 1096, 1128, 1012) | 151.32 (39.09) | 104.34 (37.09) | -28.93 (23.52)
  TG (n = 1843, 1824, 1766) | 200.07 (128.76) | 168.33 (102.82) | -7.37 (41.99)

ADVERSE EVENTS:
Time Frame: Year 1 through Year 6. There were no SAE's reported in Year three.
Groups:
- VYTORIN YEAR 1: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Year 1
- VYTORIN YEAR 2: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Year 2
- VYTORIN YEAR 4: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Year 4
- VYTORIN YEAR 5: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Year 5
- VYTORIN YEAR 6: Participants with atherosclerosis treated with Vytorin ranging from 10/10 mg/day through 10/80 mg/day for Year 6
Arm/Group | VYTORIN YEAR 1 | VYTORIN YEAR 2 | VYTORIN YEAR 4 | VYTORIN YEAR 5 | VYTORIN YEAR 6
Serious Adverse Events (participants affected / at risk) | 0/9 | 4/933 | 6/531 | 0/380 | 5/158
Other Adverse Events (participants affected / at risk) | 0/9 | 0/933 | 0/531 | 0/380 | 0/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VYTORIN YEAR 1 (N=9) | VYTORIN YEAR 2 (N=933) | VYTORIN YEAR 4 (N=531) | VYTORIN YEAR 5 (N=380) | VYTORIN YEAR 6 (N=158)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETIC FOOT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVIX CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No